CLINICAL TRIAL: NCT01996787
Title: The Clinical Performance of the Clariti Contact Lens (Including Handling Tint) for Daily Wear
Brief Title: Clinical Study of Visibility Tinted Clariti Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sauflon Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: S13-540
Record Dates: First submitted 2013-11-07; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Hyperopia; Myopia
Keywords: visibility tinted silicone hydrogel contact lenses for daily wear
MeSH Terms: conditions — Hyperopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Optix Aqua (Active Comparator): Compare safety and efficacy of the lens using OptiFree Replenish solution
  Interventions: Device: Air Optix Aqua; Device: Clariti with Handling Tint
- Clariti with Handling Tint (Active Comparator): Compare safety and efficacy of the lens using OptiFree Replenish solution
  Interventions: Device: Air Optix Aqua; Device: Clariti with Handling Tint

INTERVENTIONS:
Device: Air Optix Aqua — Lenses will be worn on a daily wear basis (i.e. removed at night and stored in solution) and worn in the normal way. Lenses will be worn for one month. Lenses should be worn for a minimum of six hours a day, four days a week. The lenses are also to be worn for a minimum of two hours before attending all follow-up visits.
Device: Clariti with Handling Tint — Lenses will be worn on a daily wear basis (i.e. removed at night and stored in solution) and worn in the normal way. Lenses will be worn for one month. Lenses should be worn for a minimum of six hours a day, four days a week. The lenses are also to be worn for a minimum of two hours before attending all follow-up visits.

SUMMARY:
The purpose of this study was to investigate the safety and efficacy of the Sauflon Clariti Monthly silicone hydrogel contact lenses with handling tint (Sauflon Pharmaceuticals Limited) by comparison with Air Optix Aqua silicone hydrogel lenses (Alcon Inc.)

Subjects used OptiFree Replenish solution (Alcon Lboratories Inc.) for daily lens maintenance, care and storage.

DETAILED DESCRIPTION:
I. Study characteristics:

The clinical study evaluates the clinical performance of a silicone hydrogel contact lens for daily wear, Clariti (including handling tint) (Sauflon Pharmaceuticals Ltd.) versus a predicate device, Air Optix Aqua (Alcon Inc.), in terms of lens performance, physiological response and subjective acceptance.

Subjects used OptiFRee Replenish solution (Alcon Laboratories Inc.) for daily lens maintenance, care and storage.

The key features were as follows:

1. One month duration.
2. Three investigator sites.
3. Daily wear soft (hydrophilic) silicone hydrogel contact lenses, replaced on a monthly basis: Clariti Monthly (with handling tint)and Air Optix Aqua. Replenish was used as a care system by all subjects.
4. A total of 38 subjects were enrolled, and 38 subjects accounted for 76 eyes were dispensed lenses. This group was randomized into 25 test subjects (50 eyes) and 13 control subjects (26 eyes).
5. Of the 25 test subjects, 25 (100%) completed one month of use. Of the 13 control subjects, 12 (92.3%)completed one month of use.
6. There were no adverse reactions.

II. Study period:

The study was conducted over one month of wear. Subjects were examined initially, and at two follow-up visits after two weeks and four weeks respectively. Study visits commenced on June 26, 2013 and completed on September 14, 2013.

ELIGIBILITY:
Inclusion Criteria:

* They are 18 years of age and above
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent
* They are willing and able to follow the protocol
* The agree not to paticipate in other clinical research for the duration of this study
* They have a best spectacle corrected visual acuity greater or equal to 20/25 (logMAR 0.1)
* They have a manifest cylinder less than or equal to 0.75D
* They have successfully worn contact lenses within six months of starting the study
* They can be fitted with spherical soft contact lenses within the power range available
* They are willing to wear the study lenses for a minimum of four days a week, six hours a day

Exclusion Criteria:

* They have any active anterior segment ocular disease which would normally contraindicate contact lens wear
* They have any anterior segment infection, inflammation or abnormality
* They use any systemic medications which would normally contraindicate contact lens wear
* They are using any ocular medications
* They have a history of herpetic keratitis
* They have a systemic disorder which would normally contraindicate contact lens wear
* They have any infectious disease (e.g. Hepatitis) or any immunosuppressive disease (e.g. HIV)
* They have glaucoma (high pressure in the eye), have had cataract surgery or a history of recurring abrasions
* They have had corneal refractive surgery or they have an irregular cornea
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus
* They are pregnant or lactating
* They have any slit lamp findings which are more serious than grade 1
* They have a history of anaphylaxis or severe allergic reactions
* They have taken part in any other contact lens or contact lens care product clinical trial or research, within two weeks prior to starting this study

Ages: 19 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Slit lamp Biomicroscopy | 1 month
  Slit Lamp examination will be performed at the initial and follow-up visits. Slit lamp findings will be graded on a 0-4 scale (0=none;4=severe).
Adverse reactions | 1 month
  Adverse reactions will be recorded throughout the study. Adverse recations will be classified as serious, significant and non-significant.
Wear Time | 1 month
  Lens wear time is recorded for the two study lenses at follow-up visits.
Visual Acuity | 1 month
  LogMAR Visual Acuity at high contrast will be recorded before and after performeing an over-refraction at the initial, two-week and one-month visits.

SECONDARY OUTCOMES:
Subjective Scores | 1 month
  Subjective scores for comfort, vision, handling and overall score will be recorded at the initial and follow-up visits. The subjective scores will be graded on a 0-5 scale.
Symptoms, problems and complaints | 1 month
  The presence or absence of symptoms, problems and complaints will be recorded at two-weeks and one-month visits.
Discontinuations | 1 month
  All subjects discontinuations will be recorded at the two-week and one-month visits.
Refraction | 1 month
  Refraction was undertaken and recorded for all subjects at the initial, two-weeks and one-month visits.
Keratometry | 1 month
  Keratometry measures will be performed at the initial and one-month visits for all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD, Principal Investigator — MCOptom FAAO FBCLA
Locations (1):
- Eurolens Research Faculty of Life Sciences The University of Manchester, Manchester, Manchester, United Kingdom

REFERENCES:
- [Result] Varikooty J, Keir N, Richter D, Jones LW, Woods C, Fonn D. Comfort response of three silicone hydrogel daily disposable contact lenses. Optom Vis Sci. 2013 Sep;90(9):945-53. doi: 10.1097/OPX.0b013e31829d8dbf. PMID 23892493
- [Result] Belda-Salmeron L, Ferrer-Blasco T, Albarran-Diego C, Madrid-Costa D, Montes-Mico R. Diurnal variations in visual performance for disposable contact lenses. Optom Vis Sci. 2013 Jul;90(7):682-90. doi: 10.1097/OPX.0b013e318299088f. PMID 23770656
- [Result] Montes-Mico R, Belda-Salmeron L, Ferrer-Blasco T, Albarran-Diego C, Garcia-Lazaro S. On-eye optical quality of daily disposable contact lenses for different wearing times. Ophthalmic Physiol Opt. 2013 Sep;33(5):581-91. doi: 10.1111/opo.12044. Epub 2013 Mar 19. PMID 23510388
- See also: Clinical Study of Clariti Monthly Contact Lens — http://clinicaltrials.gov/ct2/show/NCT01392950?term=Clariti&rank=1